CLINICAL TRIAL: NCT06527846
Title: Post Marketing Surveillance on Long Term Use of JARDIANCE® Tablets in Patients With Chronic Kidney Disease in Japan
Brief Title: Post Marketing Surveillance of JARDIANCE in Chronic Kidney Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0340
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic kidney disease (CKD)
  Interventions: Drug: JARDIANCE®

INTERVENTIONS:
Drug: JARDIANCE® — JARDIANCE®
  Other Names: Empagliflozin

SUMMARY:
Study objective is to investigate the safety and effectiveness of long-term daily use of JARDIANCE® Tablets in patients with chronic kidney disease under real-world use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD who are prescribed JARDIANCE® Tablets for CKD according to the current Japanese package insert and who provided written informed consent prior to enrolment in this study.
* Patients who have never been treated with JARDIANCE® Tablets (including treatment for Type 2 diabetes mellitus (T2DM) and/or chronic heart failure (CHF)) before enrolment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic kidney disease (CKD) who are prescribed JARDIANCE® Tablets for CKD according to the current Japanese package insert and never been treated with JARDIANCE® Tablets before enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Drug Reactions (ADRs) | Up to 52 weeks

SECONDARY OUTCOMES:
Kidney disease progression | Up to 52 weeks
  Kidney disease progression defined as incidence of end stage kidney disease (ESKD), a sustained decline in estimated glomerular filtration rate (eGFR) to <10 mL/min/1.73 m^2, renal death, or a sustained decline of ≥40% in eGFR from baseline).
  ESKD is defined as the initiation of maintenance dialysis or receipt of a kidney transplant.
Incidence of cardiovascular death | Up to 52 weeks
Incidence of all cause death | Up to 52 weeks
Incidence of hospitalization for heart failure | Up to 52 weeks
Change from baseline in eGFR to the last observation on treatment | at baseline, at last observation on treatment (Up to 52 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com